CLINICAL TRIAL: NCT02358369
Title: A Phase 2 Prospective, Multicenter, Randomized, Double-masked, Controlled Study to Evaluate the Efficacy and Safety and Dose-response of the Bimatoprost Ocular Insert (2.2 mg, 13 mg) With and Without Concomitant Artificial Tears Compared to a Placebo Ocular Insert With and Without Concomitant Timolol (0.5%) Ophthalmic Solution in Patients With Open-angle Glaucoma or Ocular Hypertension
Brief Title: Dose-Ranging Study of the Bimatoprost Ocular Insert
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ForSight Vision5, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FSV5-004
Record Dates: First submitted 2015-01-21; First posted 2015-02-09 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Primary Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 13 mg Bimatoprost Ocular Insert (Experimental): Washout + Placebo Ocular Insert in each eye for 4 to 6 weeks, followed by 13 mg Bimatoprost Ocular Insert in each eye (OU) for 12 weeks. Note: participants also self-administered placebo ophthalmic eye drops to each eye twice a day (BID) for the first 6 weeks. After 12 weeks, 13 mg Bimatoprost Ocular Insert in each eye for an additional 12 weeks.
  Interventions: Drug: Bimatoprost; Device: Placebo Ocular Insert; Drug: Placebo Eye Drops
- 2.2 mg Bimatoprost Ocular Insert (Experimental): Washout + Placebo Ocular Insert in each eye for 4 to 6 weeks, followed by 2.2 mg Bimatoprost Ocular Insert in each eye for 12 weeks. Note: participants also self-administered placebo ophthalmic eye drops in each eye twice a day for the first 6 weeks. After 12 weeks, 13 mg Bimatoprost Ocular Insert in each eye for an additional 12 weeks.
  Interventions: Drug: Bimatoprost; Device: Placebo Ocular Insert; Drug: Placebo Eye Drops
- Timolol 0.5% (Active Comparator): Washout + Placebo Ocular Insert in each eye for 4 to 6 weeks, followed by 0.5% timolol ophthalmic solution in each eye for 6 weeks. Note: participants simultaneously wore placebo ocular inserts for 12 weeks.
  After 12 weeks, 13 mg Bimatoprost Ocular Insert in each eye for an additional 12 weeks.
  Interventions: Drug: Bimatoprost; Drug: Timolol 0.5%; Device: Placebo Ocular Insert

INTERVENTIONS:
Drug: Bimatoprost — Bimatoprost sustained release Ocular Insert
Drug: Timolol 0.5% — BID drops OU, 0.5% ophthalmic solution
  Arms: Timolol 0.5%
Device: Placebo Ocular Insert — Placebo ocular insert OU.
Drug: Placebo Eye Drops — Placebo eye drops BID OU.
  Arms: 13 mg Bimatoprost Ocular Insert; 2.2 mg Bimatoprost Ocular Insert

SUMMARY:
The Bimatoprost Ocular Insert is intended to provide sustained delivery of bimatoprost to the ocular surface to lower the intraocular pressure (IOP) in patients with Open-Angle Glaucoma or Ocular Hypertension.

This study evaluated the safety and efficacy of two different doses of the Bimatoprost Ocular Insert, compared to an active control arm with timolol ophthalmic solution (0.5%).

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent
* At least 18 years of age
* Diagnosis in both eyes of either primary open-angle glaucoma (POAG) or ocular hypertension
* Best corrected-distance visual acuity score equivalent to 20/80 or better
* Stable visual field
* Central corneal thickness between 490 - 620 micrometers

Inclusion Criteria at the Randomization Visit:

("T" is defined as time and "hr" is defined as hour[s])

* IOP for each eye is ≥ 23 mm Hg at T=0 hr, ≥ 20 mm Hg at T=2 hr and T=8 hr.
* Inter-eye IOP difference of ≤ 5.0 mm Hg at T=0 hr, T=2 hr and T=8 hr.
* IOP for each eye is ≤ 30 mm Hg at T=0 hr, T=2 hr and T=8 hr.

Key Exclusion Criteria:

* Any known contraindication to prostaglandin analog (latanoprost, travoprost, bimatoprost, tafluprost) or timolol
* A cardiac or pulmonary condition that in the opinion of the Investigator would contraindicate the use of beta-blocker drops
* Cup-to-disc ratio of greater than 0.8
* Significant risk of angle closure due to pupil dilation, defined as a Shaffer classification of less than Grade 2 based on gonioscopy
* Ocular, orbital, and/or eyelid surgery of any type within the past six (6) months from screening date
* Laser surgery for glaucoma / ocular hypertension on one (1) or both eyes within the last six (6) months
* Past history of any incisional surgery for glaucoma at any time
* Past history of corneal refractive surgery
* Corneal abnormalities that would interfere with accurate IOP readings with an applanation tonometer
* Current participation in an investigational drug or device study or participation in such a study within 30 days of Screening
* Inability to adequately evaluate the retina
* Participants who will require contact lens use during the study period.
* Participants who currently have punctal occlusion
* Pregnant, lactating or of child-bearing potential and not using a medically acceptable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chen, PhD, Study Director — Allergan
Locations (10):
- United States (10):
  - Vold Vision, Fayetteville, Arkansas
  - Sall Medical Research Center, Artesia, California
  - Eye Research Foundation, Newport Beach, California
  - Clayton Eye Center, Morrow, Georgia
  - Mundorf Eye Center, Charlotte, North Carolina
  - Cornerstone Health Care, High Point, North Carolina
  - Apex Eye, Madeira, Ohio
  - University of Eye Specialists, Maryville, Tennessee
  - Total Eye Care, Memphis, Tennessee
  - R&R Eye Research, LLC, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 156 participants were enrolled and entered the washout placebo and trial-wear period. A total of 121 participants were randomized to one of three treatment groups.
Groups:
- Washout + Placebo Ocular Insert: Glaucoma medication washout and placebo ocular insert in each eye for 4 to 6 weeks prior to randomization.
- Placebo Ocular Insert + Timolol 0.5% (Period A/B): Following the washout period, timolol ophthalmic solution 0.5% twice a day in each eye plus placebo ocular insert in each eye for 6 weeks in Treatment Period A. In Treatment Period B participants continued to wear the placebo ocular inserts for 6 weeks but the eye drops were discontinued.
- 2.2 mg Bimatoprost Ocular Insert (Period A/B): Following the washout period, 2.2 mg Bimatoprost Ocular Insert in each eye plus placebo eye drops in each eye twice a day for 6 weeks in Treatment Period A. In Treatment Period B participants continued to wear the 2.2 mg Bimatoprost Ocular Inserts for 6 weeks but the eye drops were discontinued.
- 13 mg Bimatoprost Ocular Insert (Period A/B): Following the washout period, 13 mg Bimatoprost Ocular Insert in each eye plus placebo eye drops to each eye twice a day for 6 weeks in Treatment Period A. In Treatment Period B participants continued to wear the 13 mg Bimatoprost Ocular Inserts for 6 weeks but the eye drops were discontinued.
- 13 mg Bimatoprost Ocular Insert (Period C): Following Treatment Period A/B, 13 mg Bimatoprost Ocular Insert for 12 weeks in Period C (Week 12 to 24).
Period: Pre-Randomization Washout Period
Arm/Group | Washout + Placebo Ocular Insert | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period C)
Started | 156 | 0 | 0 | 0 | 0
Completed | 121 | 0 | 0 | 0 | 0
Not Completed | 35 | 0 | 0 | 0 | 0
Not completed — Not Qualified for Randomization | 35 | 0 | 0 | 0 | 0
Period: Treatment Period A/B
Arm/Group | Washout + Placebo Ocular Insert | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period C)
Started | 0 | 40 | 40 | 41 | 0
Completed | 0 | 38 | 38 | 37 | 0
Not Completed | 0 | 2 | 2 | 4 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 2 | 0
Period: Treatment Period C
Arm/Group | Washout + Placebo Ocular Insert | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period C)
Started | 0 | 0 | 0 | 0 | 113
Completed | 0 | 0 | 0 | 0 | 106
Not Completed | 0 | 0 | 0 | 0 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized, treated and returned for at least one post-treatment visit.
Groups:
- Placebo Ocular Insert + Timolol 0.5%: Following the washout period, timolol ophthalmic solution 0.5% twice a day in each eye plus placebo ocular inserts in each eye for 6 weeks in Treatment Period A. In Treatment Period B participants continued to wear the placebo ocular inserts for 6 weeks but the eye drops were discontinued. In Treatment Period C all participants were fitted with 13 mg Bimatoprost Ocular Inserts for 12 weeks.
- 2.2 mg Bimatoprost Ocular Insert: Following the washout period, 2.2 mg Bimatoprost Ocular Insert in each eye plus placebo eye drops in each eye twice a day for 6 weeks in Treatment Period A. In Treatment Period B participants continued to wear the 2.2 mg Bimatoprost Ocular Inserts for 6 weeks but the eye drops were discontinued. In Treatment Period C all participants were fitted with 13 mg Bimatoprost Ocular Insert in each eye for 12 weeks.
- 13 mg Bimatoprost Ocular Insert: Following the washout period, 13 mg Bimatoprost Ocular Insert in each eye plus placebo eye drops in each eye twice a day for 6 weeks in Treatment Period A. In Treatment Period B participants continued to wear the 13 mg Bimatoprost Ocular Inserts for 6 weeks but the eye drops were discontinued. In Treatment Period C all participants were fitted with 13 mg Bimatoprost Ocular Insert in each eye for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo Ocular Insert + Timolol 0.5% | 2.2 mg Bimatoprost Ocular Insert | 13 mg Bimatoprost Ocular Insert | Total
Number analyzed (Participants) | 40 | 40 | 41 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.70) | 64.1 (9.24) | 63.0 (10.01) | 64.9 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 20 | 35 | 82
  Male | 13 | 20 | 6 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure (IOP) at Week 8
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (T=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Week 8. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated an improvement.
Time Frame: Baseline (Day 0) to Week 8
Population: Participants from the FAS, all participants who were randomized, treated and returned for at least one post-treatment visit, with data available at Week 8.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B)
Number analyzed (Participants) | 38 | 35 | 36
mm Hg
  Change from Baseline to Week 8 (T=0 hour) | -4.68 (2.931) | -3.68 (3.105) | -4.56 (3.007)
  Change from Baseline to Week 8 (T=2 hour) | -3.62 (2.924) | -3.31 (3.063) | -3.98 (3.522)
  Change from Baseline to Week 8 (T=8 hour) | -3.21 (2.812) | -3.23 (2.573) | -3.22 (3.061)

2. Primary Outcome: Change From Baseline in IOP at Week 12
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (T=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Week 12. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated an improvement.
Time Frame: Baseline (Day 0) to Week 12
Population: FAS, all participants who were randomized, treated and returned for at least one post-treatment visit, with data available at Week 12. Participants on rescue therapy with missing data during the evaluation period or measurements out of the pre-specified visit window had IOP data imputed using LOCF (last observation carried forward) for the visit.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B)
Number analyzed (Participants) | 38 | 35 | 37
mm Hg
  Change from Baseline to Week 12 (T=0 hour) | -3.37 (3.147) | -3.64 (3.454) | -4.08 (2.893)
  Change from Baseline to Week 12 (T=2 hour) | -2.74 (2.891) | -3.67 (3.182) | -3.40 (3.815)
  Change from Baseline to Week 12 (T=8 hour) | -2.34 (2.756) | -3.20 (2.491) | -2.69 (2.523)

3. Primary Outcome: Percentage of Participants by Change From Baseline in Best-corrected Visual Acuity (BCVA) Categories at Week 8
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Time Frame: Baseline (Day 0) to Week 8
Population: Participants from the Safety Population, all randomized participants who had an ocular insert placed, with data available for analysis at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B)
Number analyzed (Participants) | 38 | 39 | 36
percentage of participants
  Right Eye, 10+ Letter Improvement | 2.6 | 0 | 2.8
  Right Eye, 5+ Letter Improvement | 18.4 | 7.7 | 5.6
  Right Eye, No Change | 65.8 | 69.2 | 77.8
  Right Eye, 5- Letter Worsening | 13.2 | 17.9 | 13.9
  Right Eye, 10- Letter Worsening | 0 | 5.1 | 0
  Left Eye, 10+ Letter Improvement | 2.6 | 0 | 5.6
  Left Eye, 5+ Letter Improvement | 10.5 | 20.5 | 19.4
  Left Eye, No Change | 68.4 | 66.7 | 66.7
  Left Eye, 5- Letter Worsening | 15.8 | 7.7 | 5.6
  Left Eye, 10- Letter Worsening | 2.6 | 5.1 | 2.8

4. Primary Outcome: Percentage of Participants by Change From Baseline in Best-corrected Visual Acuity (BCVA) Categories at Week 12
Description: as for outcome 3
Time Frame: Baseline (Day 0) to Week 12
Population: Participants from the Safety Population, all randomized participants who had an ocular insert placed, with data available for analysis at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B)
Number analyzed (Participants) | 38 | 38 | 36
percentage of participants
  Right Eye, 10+ Letter Improvement | 0 | 0 | 2.8
  Right Eye, 5+ Letter Improvement | 7.9 | 5.3 | 11.1
  Right Eye, No Change | 73.7 | 57.9 | 61.1
  Right Eye, 5- Letter Worsening | 13.2 | 28.9 | 22.2
  Right Eye, 10- Letter Worsening | 5.3 | 7.9 | 2.8
  Left Eye, 10+ Letter Improvement | 0 | 0 | 5.6
  Left Eye, 5+ Letter Improvement | 7.9 | 13.2 | 19.4
  Left Eye, No Change | 71.1 | 68.4 | 61.1
  Left Eye, 5- Letter Worsening | 18.4 | 15.8 | 13.9
  Left Eye, 10- Letter Worsening | 2.6 | 2.6 | 0

5. Primary Outcome: Percentage of Participants With Clinically Significant Change From Baseline in Slit-Lamp Examination Findings at Week 12
Description: The clinician examined and graded the eyelids, conjunctiva, cornea and anterior chamber of the eye with the aid of a slit-lamp, (conjunctival erythema was assessed as part of the examination). Fluorescein dye was instilled into the ocular cul-de-sac to facilitate this examination.
Time Frame: Baseline (Day 0) to Week 12
Population: Safety population included all participants who had an ocular insert placed.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B)
Number analyzed (Participants) | 40 | 40 | 41
percentage of participants | 0 | 0 | 0

6. Primary Outcome: Change From Baseline in Automated Visual Field at Week 12
Description: Automated Visual Field was examined used the Humphrey Visual Field Analyzer, a test that measures the entire area of peripheral vision that can be seen while the eye is focused on a central point. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 12
Population: Safety Population included all randomized participants who had an ocular insert placed. The number of participants analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: decibels (dB)
Arm/Group | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B)
Number analyzed (Participants) | 40 | 40 | 41
decibels (dB)
  Baseline | -2.58 (3.377) | -1.45 (4.041) | -2.70 (2.934)
  Change from Baseline to Week 12: number analyzed (Participants) | 38 | 38 | 36
  Change from Baseline to Week 12 | -0.18 (2.010) | 0.02 (1.819) | 0.39 (1.446)

7. Primary Outcome: Dilated Fundus Exam: Cup-to-Disc-Ratio
Description: The cup-to-disk-ratio is an eye test to assess the progression of glaucoma. The diameter of the cup is compared to the diameter of the disk and a ratio is determined. The normal cup-disk ratio is 0.3. An increase in the cup-to-disc-ratio is a possible indication of glaucoma.
Time Frame: Week 12
Population: Participants from the Safety Population, all randomized participants who had an ocular insert placed, with data available for analysis. The number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B)
Number analyzed (Participants) | 38 | 38 | 36
ratio
  Right Eye, Week 12 | 0.53 (0.172) | 0.55 (0.161) | 0.47 (0.184)
  Left Eye, Week 12 | 0.54 (0.160) | 0.56 (0.157) | 0.48 (0.176)

8. Primary Outcome: Percentage of Participants by Dilated Fundus Exam Pathology Grade at Week 12
Description: Dilated fundus examination pathology findings were noted, described and graded on a scale of None (0), Mild (+1), Moderate (+2) and Severe (+3). The percentage of participants in each grade is reported.
Time Frame: Week 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B)
Number analyzed (Participants) | 40 | 40 | 41
percentage of participants
  Right Eye, None: number analyzed (Participants) | 38 | 38 | 36
  Right Eye, None | 63.2 | 71.1 | 50.0
  Left Eye, None: number analyzed (Participants) | 37 | 38 | 36
  Left Eye, None | 62.2 | 71.1 | 47.2
  Right Eye, Mild: number analyzed (Participants) | 38 | 38 | 36
  Right Eye, Mild | 34.2 | 26.3 | 44.4
  Left Eye, Mild: number analyzed (Participants) | 37 | 38 | 36
  Left Eye, Mild | 35.1 | 26.3 | 50.0
  Right Eye, Moderate: number analyzed (Participants) | 38 | 38 | 36
  Right Eye, Moderate | 2.6 | 2.6 | 5.6
  Left Eye, Moderate: number analyzed (Participants) | 37 | 38 | 36
  Left Eye, Moderate | 2.7 | 2.6 | 2.8

9. Primary Outcome: Percentage of Participants With Ocular and Non-ocular Adverse Events (AE) by Severity in Period A/B
Description: An AE was defined as any untoward medical occurrence (eg, sign, symptom, disease, syndrome, intercurrent illness) that occurred in a study participant, regardless of the suspected cause during the study. An ocular AE is an AE that occurred in the eye and non-ocular is an AE that occurred not in the eye. Th investigator assessed the worst severity of each AE as: Mild=aware of sign or symptom, but readily tolerated, Moderate=discomfort enough to cause interference with usual activity or Severe=incapacitating with inability to work or do usual activity.
Time Frame: Baseline (Day 0) to Week 12
Population: Safety Population included all randomized participants who had an ocular insert placed.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B)
Number analyzed (Participants) | 40 | 40 | 41
percentage of participants
  Ocular, Mild | 12.5 | 17.5 | 26.8
  Ocular, Moderate | 2.5 | 5.0 | 4.9
  Ocular, Severe | 0 | 0 | 0
  Non-ocular, Mild | 5.0 | 5.0 | 9.8
  Non-Ocular, Moderate | 15.0 | 2.5 | 7.3
  Non-ocular, Severe | 0 | 2.5 | 0

10. Primary Outcome: Percentage of Participants With Ocular and Non-ocular Adverse Events (AE) by Severity in Period C
Description: An AE was defined as any untoward medical occurrence (eg, sign, symptom, disease, syndrome, intercurrent illness) that occurred in a study participant, regardless of the suspected cause during the study. An ocular AE is an AE that occurred in the eye and non-ocular is an AE that occurred not in the eye. The investigator assessed the worst severity of each AE as: Mild=aware of sign or symptom, but readily tolerated, Moderate=discomfort enough to cause interference with usual activity or Severe=incapacitating with inability to work or do usual activity.
Time Frame: Week 12 to Week 24
Population: Safety Population included all randomized participants who had an ocular insert placed.
Measure: Number; unit: percentage of participants
Groups:
- 13 mg Bimatoprost Ocular Insert (Period C): Following Treatment Period A/B, 13 mg Bimatoprost Ocular Insert in each eye for 12 weeks in Period C (Week 12 to Week 24).
Arm/Group | 13 mg Bimatoprost Ocular Insert (Period C)
Number analyzed (Participants) | 113
percentage of participants
  Ocular, Mild | 23.9
  Ocular, Moderate | 5.3
  Ocular, Severe | 0
  Non-ocular, Mild | 5.3
  Non-ocular, Moderate | 4.4
  Non-ocular, Severe | 0.9

11. Secondary Outcome: Change From Baseline in IOP at Week 2
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (T=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Week 2. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated an improvement.
Time Frame: Baseline (Day 0) to Week 2
Population: Participants from the FAS, all participants who were randomized, treated and returned for at least one post-treatment visit, with data available at Week 2.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B)
Number analyzed (Participants) | 39 | 40 | 40
mm Hg
  Change from Baseline to Week 2 (T=0 hour) | -6.84 (2.264) | -4.56 (3.134) | -5.95 (2.367)
  Change from Baseline to Week 2 (T=2 hour): number analyzed (Participants) | 39 | 40 | 39
  Change from Baseline to Week 2 (T=2 hour) | -5.71 (2.277) | -4.14 (2.637) | -5.34 (2.499)
  Change from Baseline to Week 2 (T=8 hour): number analyzed (Participants) | 39 | 40 | 38
  Change from Baseline to Week 2 (T=8 hour) | -4.81 (2.612) | -3.76 (2.320) | -4.52 (2.594)

12. Secondary Outcome: Change From Baseline in IOP at Week 6
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (T=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Week 6. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated an improvement.
Time Frame: Baseline (Day 0) to Week 6
Population: Participants from the FAS, all participants who were randomized, treated and returned for at least one post-treatment visit, with data available at Week 6.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo Ocular Insert + Timolol 0.5% (Period A/B) | 2.2 mg Bimatoprost Ocular Insert (Period A/B) | 13 mg Bimatoprost Ocular Insert (Period A/B)
Number analyzed (Participants) | 39 | 36 | 38
mm Hg
  Change from Baseline to Week 6 (T=0 hour) | -6.42 (2.770) | -4.87 (3.212) | -5.30 (2.941)
  Change from Baseline to Week 6 (T=2 hour): number analyzed (Participants) | 38 | 36 | 38
  Change from Baseline to Week 6 (T=2 hour) | -4.97 (2.948) | -4.40 (3.138) | -4.42 (2.830)
  Change from Baseline to Week 6 (T=8 hour): number analyzed (Participants) | 38 | 36 | 38
  Change from Baseline to Week 6 (T=8 hour) | -4.40 (2.529) | -3.73 (2.393) | -3.77 (2.291)

13. Secondary Outcome: Change From Baseline in IOP in Period C
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (T=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Weeks 14, 18 and 24. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal timepoint. A negative change from Baseline indicated an improvement.
Time Frame: Baseline (Day 0) to Weeks 14, 18 and 24
Population: Participants from the FAS, all participants who were randomized, treated and returned for at least one post-treatment visit, with data available at the given timepoint.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | 13 mg Bimatoprost Ocular Insert (Period C)
Number analyzed (Participants) | 113
mm Hg
  Change from Baseline to Week 14 (T=0 hour): number analyzed (Participants) | 101
  Change from Baseline to Week 14 (T=0 hour) | -5.72 (2.919)
  Change from Baseline to Week 14 (T=2 hour): number analyzed (Participants) | 101
  Change from Baseline to Week 14 (T=2 hour) | -4.64 (3.100)
  Change from Baseline to Week 14 (T=8 hour): number analyzed (Participants) | 101
  Change from Baseline to Week 14 (T=8 hour) | -4.13 (2.849)
  Change from Baseline to Week 18 (T=0 hour): number analyzed (Participants) | 98
  Change from Baseline to Week 18 (T=0 hour) | -5.62 (3.135)
  Change from Baseline to Week 18 (T=2 hour): number analyzed (Participants) | 98
  Change from Baseline to Week 18 (T=2 hour) | -4.33 (3.072)
  Change from Baseline to Week 18 (T=8 hour): number analyzed (Participants) | 98
  Change from Baseline to Week 18 (T=8 hour) | -4.17 (2.714)
  Change from Baseline to Week 24 (T=0 hour): number analyzed (Participants) | 93
  Change from Baseline to Week 24 (T=0 hour) | -4.85 (2.882)
  Change from Baseline to Week 24 (T=2 hour): number analyzed (Participants) | 93
  Change from Baseline to Week 24 (T=2 hour) | -3.99 (2.847)
  Change from Baseline to Week 24 (T=8 hour): number analyzed (Participants) | 93
  Change from Baseline to Week 24 (T=8 hour) | -2.99 (3.010)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for a period of 28 to 30 weeks, from the beginning of the Washout Period (starting on Week -6 to -4) to the end of study (Week 24).
Description: During the Washout Period (4 to 6 weeks) prior to randomization, adverse event data were collected for all participants in a single arm.
  During the entire 24 weeks of treatment (consisting of Treatment Periods A, B and C), adverse event data were not collected by the intervention received, but instead, according to the arm participants were randomized to at the start of Treatment Period A (Week 0).
Arm/Group | Washout + Placebo Ocular Insert | Placebo Ocular Insert + Timolol 0.5% | 2.2 mg Bimatoprost Ocular Insert | 13 mg Bimatoprost Ocular Insert
Serious Adverse Events (participants affected / at risk) | 0/156 | 3/40 | 1/40 | 1/41
Other Adverse Events (participants affected / at risk) | 9/156 | 16/40 | 12/40 | 20/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Washout + Placebo Ocular Insert (N=156) | Placebo Ocular Insert + Timolol 0.5% (N=40) | 2.2 mg Bimatoprost Ocular Insert (N=40) | 13 mg Bimatoprost Ocular Insert (N=41)
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Device dislocation (General disorders) | 0 | 1 | 0 | 0
Brain hypoxia (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Washout + Placebo Ocular Insert (N=156) | Placebo Ocular Insert + Timolol 0.5% (N=40) | 2.2 mg Bimatoprost Ocular Insert (N=40) | 13 mg Bimatoprost Ocular Insert (N=41)
Conjunctival hyperaemia (Eye disorders) | 3 | 2 | 3 | 3
Eye discharge (Eye disorders) | 5 | 5 | 7 | 7
Eye pruritus (Eye disorders) | 1 | 3 | 2 | 1
Punctate keratitis (Eye disorders) | 0 | 3 | 1 | 6
Conjunctival haemorrhage (Eye disorders) | 0 | 2 | 2 | 1
Eye irritation (Eye disorders) | 0 | 2 | 1 | 0
Dry eye (Eye disorders) | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Hypertension (Vascular disorders) | 1 | 2 | 0 | 3
Vision blurred (Eye disorders) | 0 | 1 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No presentation or publication of Institution's data relating to the Trial may occur until after the Trial has been completed at all sites. If Investigator desires to present or publish, investigator must submit any and all manuscripts, posters, abstracts, or other intended publications (hereinafter collectively referred to as "manuscripts") to Sponsor at least sixty (60) days prior to the actual submission of such manuscript(s) for publication.